CLINICAL TRIAL: NCT02113306
Title: Does Transcutaneous Vagal Nerve Stimulation Improves Fear Extinction in Humans
Acronym: t-VNSext
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Ilse Van Diest, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: t-VNS extinction
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- t-VNS (Experimental): electrical stimulation of the concha of the ear
  30sec trains of 0.25msec-duration monophasic square wave pulses at 25Hz, with a stimulation intensity not exceeding 0.5 mA
  Interventions: Device: t-VNS
- sham t-VNS (Sham Comparator): Sham stimulation of the earlobe will be conducted by positioning the electrode upside down
  30sec trains of 0.25msec-duration monophasic square wave pulses at 25Hz, with a stimulation intensity not exceeding 0.5 mA
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: t-VNS — The device that will be used is approved for systematic use by those with epilepsy and depression in the European Union. It has been used in studies of acute stimulation with healthy participants with no significant changes in heart rate or breathing (Kraus et al., 2007; Busch et al., 2013).
  Other Names: NEMOS®, Cerbomed, Erlangen, Germany
  Arms: t-VNS
Device: sham stimulation — electrodes will be put upside down
  Other Names: NEMOS®, Cerbomed, Erlangen, Germany
  Arms: sham t-VNS

SUMMARY:
A recent study with rats showed that electrical stimulation of the vagus nerve (VNS) facilitates extinction of fear (Pena, Engineer, & McIntyre, Biological Psychiatry, 2013). The hypothesized mechanism is that VNS both enhances memory consolidation (by increasing noradrenergic neurotransmission) and reduces anxiety (thus: preventing fear responses to the CS which may re-consolidate the fear memory). The effect was only apparent when VNS occurred during exposure of the fear conditioned stimulus (CS), and not when stimulation was given immediately following exposure. These results may have implications for the treatment of anxiety disorders in humans. However, until recently, the only means to investigate the effects of VNS on human fear learning would have required the invasive implantation of vagus nerve stimulators. This has fortunately changed, as a non-invasive transcutaneous VNS device has been approved for use in the E.U. for the treatment of psychological disorders.

This study proposes to use a t-VNS to investigate its effects on fear learning and extinction in (healthy) humans. Previous research has only investigated the effects it has on human mood and memory. The results obtained suggest that it reduces negative affect and enhances memory, findings which are consistent with those reported for rats. It is thus reasonable to expect that t-VNS will facilitate the extinction of fear in humans.

The present study aims to answer the following research questions:

Does t-VNS during extinction training:

1. accelerates extinction curves
2. reduces spontaneous recovery of previously extinguished fear
3. reduce re-acquisition of fear
4. reduce generalization of fear to other stimuli that resemble the CS+?
5. facilitates the generalization of inhibitory learning to stimuli that resemble the CS-?

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women aged 16 - 50 years

Exclusion Criteria:

* current or past psychiatric or neurological disorder
* use of psychopharmaca
* use of medication that affects autonomic nervous functioning (e.g., bèta-blockers)
* current cardiac or respiratory disorder
* pregnancy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
fear response | 3 test days
  startle blink EMG skin conductance response ECG respiration self-reports

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Van Diest, PhD, Principal Investigator — KU Leuven
Locations (1):
- Faculty of Psychology and Educational Science, Leuven, Belgium